CLINICAL TRIAL: NCT01781273
Title: MedDrive's Responsiveness to Different Blood Alcohol Concentrations and Concurrent Validity Against Performances on a Driving Simulator; a Phase I, Randomised, Double Blind, Placebo, Dose Response Validation Trial
Brief Title: MedDrive's Responsiveness to Alcohol
Acronym: OH-MedDrive
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lausanne (Other)
Collaborators: University of Lausanne Hospitals (Other); University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Bernard Favrat, MD, Head of Unit of Traffic Medicine and Psychology, Principle Investigator, University of Lausanne
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Diagnostic
Other Study IDs: CE-12-277
Record Dates: First submitted 2013-01-28; First posted 2013-01-31 (Estimated); Last update posted 2013-04-23 (Estimated); Status verified 2013-04

CONDITIONS: Impaired Driving
Keywords: impaired driving
MeSH Terms: interventions — Ethanol

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Cranberry juice alone (Placebo Comparator): 500 mL of cranberry juice
  Interventions: Other: Cranberry juice
- BAC 0.5 g/L (Experimental): Cranberry juice with ethanol to rise BAC to 0.5 g/L
  Interventions: Other: Ethanol; Other: Cranberry juice
- BAC 0.65 g/L (Experimental): Cranberry juice with ethanol to rise BAC to 0.65 g/L
  Interventions: Other: Ethanol; Other: Cranberry juice
- BAC 0.8 g/L (Experimental): Cranberry juice with ethanol to rise BAC to 0.8 g/L
  Interventions: Other: Ethanol; Other: Cranberry juice

INTERVENTIONS:
Other: Ethanol — During a 45 min period, investigators will ask participants to drink 500ml of cranberry juice, 100 ml at a time each 5 minutes. Depending of the allocation, these drinks will contain more or less alcohol. Pure ethanol will be used mixed with the beverage. The amount of alcohol to dilute in the drink will be calculated using Widmarks formula. Participants will move to the simulator room 20 minutes after having finished drinking the first 500 ml. To maintain the BAC level, investigators will use a breathalyser and provide 100 ml cranberry juice every 20 minutes with the amount of necessary alcohol. The person administrating drinks will hand over the drinks and make sure the participants breaths in before taking a sip, thereby inhaling alcohol vapour from the lid and keeping them blinded to the content.
  Arms: BAC 0.5 g/L; BAC 0.65 g/L; BAC 0.8 g/L
Other: Cranberry juice — 100 mL cranberry juice is provided in a 250 ml container.

SUMMARY:
This four-way, dose-response, crossover, double blind, placebo-controlled, randomised validation study investigates the responsiveness of MedDrive, a computed battery of neuropsychological tasks, to different doses of alcohol.

The following hypothesis are tested:

1. Measures from MedDrive are influenced by alcohol in a dose dependent way.
2. Effects of alcohol on driving performances are correlated to measures from MedDrive in a dose dependent way.
3. Within a group of healthy young drivers, MedDrive shows consistent results over repeated measures (ICC≥0.7).
4. MedDrive models effects of alcohol on driving performances better than does the UFOV or the trial making task.

DETAILED DESCRIPTION:
Background: There is an increasing need for physicians to advice patients on their fitness to drive. Current guidelines underline the limitations of existing instruments and the poor adaptability of batteries of neuropsychological tests assessing fitness to drive in both experimental and primary care settings. The investigators therefore developed MedDrive, a free, reliable, computer based measuring instrument capable of detecting effects of age and drugs on cognitive functions considered as essential for driving.

Objectives: This study aims to test MedDrive responsiveness to different blood alcohol concentrations (BAC) and validate these measures against performances on a driving simulator. It also aims to measure MedDrive's reliability following repeated measures during the training phase, to compare MedDrive's performances in measuring effects of different BAC against the UFOV, and to model MedDrives measures to predict behaviour on the simulator. Finally, this study also includes a nested experimental study measuring effects of alcohol on attention.

Methods: Using Widmark's formula, 16 healthy young drivers are given cranberry juice with different doses of ethanol to bring their BAC to 0 g/L, 0.5 g/L, 0.65 g/L, and 0.8 g/L. They are blinded to the presence of ethanol by inhaling vapors of ethanol just before drinking. BAC is maintained during the entire experiment by using a breathalyser and administrating drinks throughout the experiment. Three scenarios are planned on a driving simulator (StSoftware PvW-2010), a road tracking task, a car following task, and a car following task including dual tasking using peripheral vision.

ELIGIBILITY:
Inclusion Criteria:

* Aged 20 to 40 years
* Obtained drivers license at least 24 months before
* Fit to drive
* Consumed at least once six units of a beverage with alcohol at a single occasion during the previous six months

Exclusion Criteria:

* Under the influence of a medicinal drug affecting their driving performance
* Suffer from a psychiatric condition affecting driving performances
* Suffer from simulator sickness
* Presenting criteria (ICD-10) of alcohol dependence.
* Pregnant or breastfeeding
* Intolerant to alcohol defined by having either headaches or digestive disorders for quantities of alcohol that do not seem to bother other people.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2013-02; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
central visual processing time | 1 hour post-intervention
  Corresponds to the duration of exposure in ms for a 37.5% threshold for correct guesses adjusted for chance for central vision in the Visual Recognition Task (Task 1) in MedDrive.
peripheral visual processing time | 1 hour post-intervention
  Corresponds to the duration of exposure in ms for a 43.8% threshold for correct guesses adjusted for chance for peripheral vision in the Visual Recognition Task (Task 1) in MedDrive.
dual task processing time | 1 hour post-intervention
  Corresponds to the duration of exposure in ms for a 48.7% threshold for correct guesses adjusted for chance for simultaneous central and peripheral vision (dual tasking) in the Visual Recognition Task (Task 1) in MedDrive.
neutral response time | 1 hour post-intervention
  Corresponds to the average response time in ms adjusted for learning effect for participants to respond to a peripheral stimuli during the Central Cue Attention Task (Task 2) in MedDrive.
conditioned alerting gain | 1 hour post-intervention
  Corresponds to the average gain in response time (ms) over the neutral condition after participants are warned of the imminent exposure to a peripheral stimuli during the Central Cue Attention Task (Task 2) in MedDrive.
orientation gain | 1 hour post-intervention
  Corresponds to the average gain in response time (ms) over the neutral condition after participants are shown where the peripheral stimuli is to show up during the Central Cue Attention Task (Task 2) in MedDrive.
attention shift response time | 1 hour post-intervention
  Corresponds to the average response time in ms to detect the orientation of a given moving target during the Movement Detection Task (Task 3) in MedDrive.
distance to first cue | 1 hour post-intervention
  Corresponds to the geometrical mean of distances in mm between the true location of the first cue and its indicated location during the Memory Decay of Spatial Resolution Task (Task 4) in MedDrive.
distance to last cue | 1 hour post-intervention
  Corresponds to the geometrical mean of distances in mm between the true location of the last cue and its indicated location during the Memory Decay of Spatial Resolution Task (Task 4) in MedDrive.
spatial resolution decay | 1 hour post-intervention
  Corresponds to the loss in precision for each extra cue shown during the Memory Decay of Spatial Resolution Task (Task 4) in MedDrive (ln(mm)/cue).

SECONDARY OUTCOMES:
Useful Field of View | 1 hour post-intervention
  The UFOV is a neuropsychological task which provides four outputs: visual processing, divided attention, selective attention, and overall risk
Trial Making Task | 1 hour post-intervention
  The duration of tasks TMT-A and TMT-B are provided in seconds
StSoftware driving simulator | 1 hour post-intervention
  Standard lateral deviation from the center of the road during the road tracking task, and gain and delay during the car following tasks

OTHER OUTCOMES:
Adverse events | 1 week after intervention
  New symptoms, accidents, hospitalisation are recorded one week after each visit.

CONTACTS AND LOCATIONS:
Overall Officials: Bernard Favrat, MD, Principal Investigator — CHUV, University of Lausanne; Patrice Mangin, MD, PhD, Study Director — CHUV, University of Lausanne
Locations (1):
- Institute of Legal Medicine, University of Geneva, Geneva, Canton of Geneva, Switzerland